CLINICAL TRIAL: NCT03964402
Title: Sample Size Determination in Heterogeneous Populations for Multivariate Time-to-event Data
Brief Title: Sample Size for Multivariate Time-to-event Data
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: IB2018-SAMPLE-SIZE-SURVIVAL
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Clinical Trials
Keywords: sample size, survival, randomized clinical trials, statistical test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical trial: Corresponds to a comparative clinical trial for which our new statistical methods will be applied to estimate sample size

SUMMARY:
Most of randomized clinical trials (RCT) using time-to-event criteria as the primary endpoint are designed, powered and analyzed based on an hypothetical hazard ratio (HR) corresponding to the targeted effect size between experimental and control arms. Usually, one assumes that populations are homogeneous within each treatment arm, that is, within each arm, (i) the baseline risk is identical for all patients, and (ii) the treatment effect is identical for all patients. This assumption however may not hold in all circumstances. This project aims at providing a statistical method for the estimation of sample size in RCT, in the presence of heterogenous populations, such as assuming populations with distinct underlying baseline risks or assuming different treatment effects.

ELIGIBILITY:
Any comparative clinical trial for which modern statistical methods are required to estimate sample size

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any comparative clinical trial for which modern statistical methods are required to estimate sample size, in particular, it can be clinical trials :
  * with heterogeneous populations,
  * with recurrent event data,
  * involving a biomarker-Strategy Designs With Multiple Treatments.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  time from randomization to death

CONTACTS AND LOCATIONS:
Overall Officials: Carine Bellera, PhD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Comprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinart D, Bellera C, Rondeau V. Sample size estimation for cancer randomized trials in the presence of heterogeneous populations. Biometrics. 2022 Dec;78(4):1662-1673. doi: 10.1111/biom.13527. Epub 2021 Sep 3. PMID 34242412
- [Background] Dinart D, Bellera C, Rondeau V. Sample size estimation for recurrent event data using multifrailty and multilevel survival models. J Biopharm Stat. 2025 Mar;35(2):241-256. doi: 10.1080/10543406.2024.2310306. Epub 2024 Feb 9. PMID 38334044
- [Background] Dinart D, Rondeau V, Bellera C. Sample Size Estimation Using a Partially Clustered Frailty Model for Biomarker-Strategy Designs With Multiple Treatments. Pharm Stat. 2024 Nov-Dec;23(6):1084-1094. doi: 10.1002/pst.2407. Epub 2024 Jul 16. PMID 39014905